CLINICAL TRIAL: NCT04333355
Title: Phase 1 Study to Evaluate the Safety of Convalescent Plasma as an Adjuvant Therapy in Patients With SARS-CoV-2 Infection
Brief Title: Safety in Convalescent Plasma Transfusion to COVID-19
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Other clinical trails probed that the use of convalescent plasma for patients with COVID-19 is safe .
Sponsor: TecSalud Investigación Clínica (Other)
Collaborators: Tecnologico de Monterrey (Other)
Responsible Party: Principal Investigator, Servando Cardona-Huerta, Director of Clinical Research, TecSalud Investigación Clínica
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PC-TecSalud Fase I
Record Dates: First submitted 2020-03-31; First posted 2020-04-03 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; Convalescent plasma
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID-19 patients receiving Convalescent Plasma (Experimental): Convalescent Plasma from patients who recently recover from COVID-19
  Interventions: Biological: Convalescent Plasma

INTERVENTIONS:
Biological: Convalescent Plasma — Along with the administration of convalescent plasma, patients will continue to receive supportive standard care.
  Other Names: Supportive standard care

SUMMARY:
There is currently no specific vaccine or treatment to treat critically ill patients with COVID-19. Different therapies are still under investigation and are use in different health institutions, however, a significant proportion of patients do not respond to these treatments, so it is important to seek new treatments. One of these alternatives is the use of convalescent plasma. The investigator will use plasma obtained from convalescent individuals with proven novel SARS-CoV-2 virus infection, diagnosed with coronavirus-19-induced disease and symptom-free for a period of not less than 10 days since they recovered from the disease. This plasma will be infused in patients affected by the same virus, but who have developed respiratory complications that have not responded favorably to usual treatment such as chloroquine, hydroxychloroquine, azithromycin, and other antivirals. The investigator will evaluate the safety of this procedure by accounting for any adverse event.

DETAILED DESCRIPTION:
There is currently no specific vaccine or treatment to treat critically ill patients with COVID-19. Different therapies are still under investigation and are use in different health institutions, however, a significant proportion of patients do not respond to these treatments, so it is important to seek new treatments. One of these alternatives is the use of convalescent plasma.

The investigator will use plasma obtained from convalescent individuals with proven novel SARS-CoV-2 virus infection, diagnosed with coronavirus-19-induced disease and symptom-free for a period of not less than 10 days since they recovered from the disease. Donors will be screened for infectious diseases including sARS-CoV-2 and will be programmed for apheresis the next day. The investigaotr will process one plasmatic volume per donor and this will be guarded in the blood bank until required by the principal investigator.

Patients or receptors will be screened and selected by the research team according to eligibility criteria, including severe disease refractory to treatment such as chloroquine, hydroxychloroquine, azithromycin, and other antivirals. Plasma will be fractioned in 250ml. Infusion will start after a clinical evaluation and blood sampling. Patients will remain under careful observation. If no adverse event is present, infusion will be repeated after 24 hours and the investigator will evaluate patients again 48 hours after the second transfusion. A final evaluation will be performed at day 14. The investigator will evaluate the safety of this procedure by accounting for any adverse event.

ELIGIBILITY:
Inclusion Criteria

1. Patients 18 years and older
2. Confirmed SARS-CoV-2 Infection by RT-PCR.
3. Serious or life-threatening infection defined as:

   Serious:
   1. Dyspnea
   2. Respiratory rate greater than or equal to 30 cycles / minute.
   3. Blood oxygen saturation less than or equal to 93% with an oxygen supply greater than 60%.
   4. Partial pressure of arterial oxygen to fraction of inspired oxygen ratio < 300
   5. A 50% increase in pulmonary infiltrates defined by computer tomography scans in 24 to 48 hours.

      Life-threatening infection:
   6. respiratory failure.
   7. septic shock.
   8. dysfunction or multiple organ failure.
4. Refractory to treatment with azithromycin / hydroxychloroquine or chloroquine / ritonavir / lopinavir defined as: 48 hours with no improvement in the modified parameters such as serious or clinically imminent infection.
5. Signed Informed consent by the patient or by the person responsible for the patient in the case of critically ill patients (spouse or parents).

Exclusion Criteria:

1. Patients with a history of allergic reaction to any type of previous transfusion.
2. Heart failure patients at risk of volume overload.
3. Patients with a history of chronic kidney failure in the dialysis phase.
4. Patients with previous hematological diseases (anemia less than 10 grams of hemoglobin, platelets greater than 100,000 / µl).
5. Any case where the investigator decides that the patient is not suitable for the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
Side effects | 14 days
  Identify possible adverse effects after the administration of convalescent plasma

SECONDARY OUTCOMES:
Heart Failure | 14 days
  Development of heart failure during convalescent plasma transfusion or after it.
Pulmonary Edema | 14 days
  Development of pulmonary edema during convalescent plasma transfusion or after it.
Allergic Reaction | 14 days
  Development of any allergic reaction during convalescent plasma transfusion or after it.
Viral load of SARS-CoV-2 | 48 hrs
  RT PCR SARS-CoV-2
Viral load of SARS-CoV-2 | 14 days
  RT PCR SARS-CoV-2

CONTACTS AND LOCATIONS:
Overall Officials: José Fe Castilleja-Leal, MD., Principal Investigator — Hospital San José
Locations (1):
- Hospital San José, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Casadevall A, Pirofski LA. The convalescent sera option for containing COVID-19. J Clin Invest. 2020 Apr 1;130(4):1545-1548. doi: 10.1172/JCI138003. No abstract available. PMID 32167489